CLINICAL TRIAL: NCT02755545
Title: A Multi-Center Clinical Trial to Evaluate the Efficacy of Two Acne Treatments
Brief Title: A Clinical Trial to Evaluate the Efficacy of Two Acne Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10354
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Salicylic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Product A (adapalene) (Active Comparator): Product A applied topically to the entire face or other affected area of the skin once daily
  Interventions: Drug: Product A
- Product B (salicylic acid) (Active Comparator): Product B applied topically to the affected area of the skin 1 to 3 times daily.
  Interventions: Drug: Product B

INTERVENTIONS:
Drug: Product A — Product A applied topically to the entire face or other affected area of the skin once daily
  Other Names: Adapalene
  Arms: Product A (adapalene)
Drug: Product B — Product B applied topically to affected area of the skin 1 to 3 times daily
  Other Names: Salicylic acid
  Arms: Product B (salicylic acid)

SUMMARY:
The purpose of this study is to evaluate the efficacy of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

DETAILED DESCRIPTION:
1. To characterize the effectiveness of the acne treatment in lesion count at week 1, week 2, week 6, week 12, and week 24 as compared to baseline and compare between treatments
2. To characterize the effectiveness of the acne treatment in Investigator's Global Improvement Assessment at week 1, week 2, week 6, week 12, and week 24 as compared to baseline and compare between treatments
3. To characterize the effect of the acne treatment in clinical grading of efficacy parameters through digital images at week 6, week 12, and week 24 as compared to baseline and compare between treatments
4. To characterize the effect of the acne treatment in subject self-assessment questionnaire responses at week 1, week 2, week 6, week 12, and week 24 as compared to baseline and compare between treatments

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women age 21 to 45 years at the time of enrollment.
2. Individuals with mild to moderate acne (score of 2-3 on FDA Investigator's Global Assessment Scale1) on the face.
3. Individuals with at least 5 inflammatory lesions.
4. Individuals with 10 - 100 non-inflammatory lesions.
5. Fitzpatrick skin type I-VI
6. Individuals willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and are able to read, speak,write, understand English.
7. Willing to withhold all facial treatments during the course of the study
8. Individuals of child bearing potential who use an acceptable method of contraception throughout the study.
9. Subjects must be stable on any medication they are taking for at least 30 days.

Key Exclusion Criteria:

1. Individuals diagnosed with allergies to topical acne products.
2. Individuals having a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
3. Women who are nursing, pregnant, or planning to become pregnant during the study.
4. Individuals who have pre-existing or dormant dermatologic conditions on the face which in the opinion of the Investigator could interfere with the outcome of the study.
5. Individuals using or who have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
6. Individuals who are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
7. Individuals with any planned surgeries and/or invasive medical procedures during the course of the study.
8. Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
9. Individuals with facial sunburn or excessive tanned facial skin or that are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
10. Individuals that are currently taking or have taken within the last 30 days oral or topical prescription medications for acne.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephens & Associates, Inc. Texas Research Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adapalene: Subjects who were randomized to adapalene and used it once-daily.
- Salicylic Acid: Subjects who were randomized to salicylic acid and used it as directed per the OTC monograph.
Period: Overall Study
Arm/Group | Adapalene | Salicylic Acid
Started | 62 | 65
Completed | 43 | 44
Not Completed | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Adapalene: Subjects who were randomized to adapalene
- Salicylic Acid: Subjects who were randomized to salicylic acid.
- Total: Total of all reporting groups
Arm/Group | Adapalene | Salicylic Acid | Total
Number analyzed (Participants) | 62 | 65 | 127
Age, Categorical [Count of Participants; unit: Participants] — Population: Some subjects were enrolled, but excluded from analysis as they were withdrawn from the study before drug dispensed.
  Participants
    number analyzed (Participants) | 58 | 59 | 117
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 58 | 59 | 117
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some subjects were enrolled, but excluded from analysis as they were withdrawn from the study before drug dispensed.
  Participants
    number analyzed (Participants) | 58 | 59 | 117
    Female | 49 | 56 | 105
    Male | 9 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some subjects were enrolled, but excluded from analysis as they were withdrawn from the study before drug dispensed.
  Participants
    number analyzed (Participants) | 58 | 59 | 117
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 24 | 24 | 48
    White | 26 | 24 | 50
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 62 | 65 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Lesions at Week 12
Description: Percent change from baseline in total lesions at week 12 was assessed by investigator or designee. Investigator or designee counted and recorded the number of open comedones, closed comedones, papules, and pustules on each subject's face. Lesions were counted globally on the following facial locations/quadrants: forehead, left cheek, chin, and right cheek. Each of the following lesion types were analyzed separately for forehead, left cheek, chin, right cheek, and the total of the 4 areas:
  * Inflammatory acne lesions (sum of papules and pustules)
  * Non-inflammatory acne lesions (sum of open comedones and closed comedones)
  * Total lesion counts (sum of inflammatory and non-inflammatory acne lesions counts)
Time Frame: Baseline and 12 weeks
Population: A total of 127 were enrolled, but only 117 were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Percent change in lesions
Groups:
- Adapalene: Subjects treated with adapalene.
- Salicylic Acid: Subjects treated with salicylic acid.
Arm/Group | Adapalene | Salicylic Acid
Number analyzed (Participants) | 58 | 59
Percent change in lesions
  Open comedones: number analyzed (Participants) | 52 | 52
  Open comedones | -17.1 (117.4) | -45.6 (61.1)
  Closed comedones: number analyzed (Participants) | 53 | 59
  Closed comedones | -13.0 (165.5) | 7.6 (153.8)
  Papules | -4.2 (71.7) | 6.4 (83.5)
  Pustules: number analyzed (Participants) | 32 | 31
  Pustules | -30.1 (153.2) | -18.2 (113.5)
  Inflammatory acne lesions | -10.0 (67.0) | 1.1 (72.6)
  Non-inflammatory acne lesions | -34.7 (41.8) | -22.8 (43.0)
  Total lesion counts | -28.3 (38.2) | -17.5 (36.7)

ADVERSE EVENTS:
Time Frame: Collected over the duration of the study up to 24 weeks.
Arm/Group | Adapalene | Salicylic Acid
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/65
Other Adverse Events (participants affected / at risk) | 2/62 | 0/65
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene (N=62) | Salicylic Acid (N=65)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02755545/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT02755545/SAP_001.pdf
  • Informed Consent Form (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT02755545/ICF_002.pdf